CLINICAL TRIAL: NCT07203651
Title: Comparison Between Diclofenac and Sterile Water Injection for Relief of Labour Associated Bachache
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Sidra Rauf, Postgraduate resident, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pakistan Institute of Medical
Record Dates: First submitted 2025-06-22; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Labour Analgesia
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group receiving intradermal sterile water injection (Experimental)
  Interventions: Drug: Sterile Water Injection
- Group receiving diclofenac injection (Experimental)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Sterile Water Injection — WE will compare effectiveness of intradermal sterile water injection with intramuscular diclofenal
  Arms: group receiving intradermal sterile water injection
Drug: Diclofenac — comparing effectiveness of diclofenac with intradermal sterile water injection
  Arms: Group receiving diclofenac injection

SUMMARY:
Comparison of Intradermal sterile water injection with diclofenac for relief of labour associated bachache

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females in active stage of labour

Exclusion Criteria:

* females asking for epidural

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant females
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 6 months
  relief of labour associated bachache using visual analogue pain scale. Scale is from 0 to 10 score. Score 0 means no pain and Score 10 keans worst possible pain.
  1-2 Score: Mild pain 3-4 score: moderate pain 5-6 score: severe pain 7-8 score: very severe 9-10: worst pain possible Having lower scores means better outcome in terms of pain relief

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided